CLINICAL TRIAL: NCT00756483
Title: Study the Effects of Pre- and Post-Operative Resistive Exercise in Total Arthroplasty Patients Using the Stability Plus Exercise System
Brief Title: Stability Plus - Outcomes From Extended Continuum of Care
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Stability Plus, LLC (Industry)
Collaborators: University of Missouri-Columbia (Other)
Responsible Party: James Yost/CEO, Stability Plus, LLC
Other Study IDs: 1107957-UMC
Record Dates: First submitted 2008-09-18; First posted 2008-09-22 (Estimated); Last update posted 2008-09-22 (Estimated); Status verified 2008-09

CONDITIONS: Arthroplasty
Keywords: Resistance; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- M, 1: Male patients that have undergone total knee replacement
- F, 1: Female patients that have undergone total knee replacement
- M, 2: Male patients that have undergone total hip replacement
- F, 2: Female patients that have undergone total hip replacement

SUMMARY:
Basic Protocol

1. Identify participant(s)
2. Request patient participation/Acquire Consent
3. Register patient at www.stabilityplus.net through the LOGIN tab

   * Patient ID (Name/Initials/SSN or any combination thereof)
   * Gender
   * Age
   * Surgical Procedure
   * Date of Surgery
   * Select Basic Exercise Program that corresponds with Surgical Procedure
4. Perform Initial Assessment using Basic Exercises for the Surgical Procedure
5. Enter Assessment Data at www.stabilityplus.net (through the LOGIN tab/Portal)
6. Within portal, modify Basic Exercise Program to create customized Stability Plus prescription for the patient
7. Monitor patient progress through Stability Plus portal.

ELIGIBILITY:
Inclusion Criteria:

* Undergone total joint replacement
* Must be able to complete pre-operative strength assessment
* Must be able to exercise using specified resistive bands

Exclusion Criteria:

* Non-ambulatory patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients that have undergone total joint replacement - hip or knee
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-03 (Estimated); Study Completion 2009-10 (Estimated)

PRIMARY OUTCOMES:
Pre- and post- study strength assessment tests for joint specific exercises | 3 months, 6 months and 12 months

SECONDARY OUTCOMES:
Reduced recovery time versus current norm | 3 months, 6 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: James T Yost, Study Director — Stability Plus, LLC
Locations (1):
- University of Missouri Hospital, Columbia, Missouri, United States